CLINICAL TRIAL: NCT06004375
Title: THE EFFECT OF ARGININE AND GLUTAMINE ON COVID-19 PATIENTS OUTCOME: A RANDOMIZED CLINICAL TRIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitas Sriwijaya (Other)
Collaborators: M. Djamil General Hospital (Unknown)
Responsible Party: Principal Investigator, Sari Bema Ramdika, Ms, Universitas Sriwijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID
Record Dates: First submitted 2023-08-19; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
Keywords: COVID-19; Oral Nutrition Supplement
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group was given a High-Calorie High-Protein + ONS diet containing 4.8 g arginine and 2 g glutamine, namely Neomune 2x 200 cc, purchased from Otsuka Pharmaceutical Co., Ltd
  Interventions: Dietary Supplement: Neomune
- control group (Active Comparator): the control was administered with a High-Calorie High-Protein diet + ONS hospital standard.
  Interventions: Dietary Supplement: Neomune

INTERVENTIONS:
Dietary Supplement: Neomune — Neomune containing 4.8 g arginine and 2 g glutamine

SUMMARY:
The goal of this clinical trial is to determine effect of arginine and glutamine on outcome of COVID-19 patients. The main questions it aims to answer are:

-to test the effect of oral nutritional supplements containing arginine and glutamine on covid-19 patients outcome Dr. M. Djamil General Hospital Padang

Participants will given ONS containing arginine and glutamine. Researchers will compare intervention group with control group to see if ONS affected outcome of COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients confirmed positive for COVID-19
* Age over 17 years
* The patient can take food orally

Exclusion Criteria:

* Patients with restricted fluid intake
* Patients who cannot take food orally
* suffering from diabetes mellitus and kidney failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
length of stay | 3 months
  length of stay of patients in hospital
Outcome | 3 months
  Outcome Measures of patients (discharge or dead)
ICU Admission | 3 months
  A patient is likely to be admitted to ICU during intervention period

SECONDARY OUTCOMES:
Il-6 and CRP Levels | 3 months
  Il-6 and CRP Levels during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. M. Djamil General Hospital, Padang, West Sumatera, Indonesia

IPD SHARING:
Plan to Share IPD: No